CLINICAL TRIAL: NCT05149118
Title: Early Postoperative Injections of Polydeoxyribonucleotide Prevents Hypertrophic Scarring After Thyroidectomy: A Randomized Controlled Trial
Brief Title: Effect of PDRN in Post-operative Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Shin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B-1811-507-005
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix | interventions — Polydeoxyribonucleotides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDRN injected group (Experimental): The participants in treatment group had received two consecutive injections of PDRN one day and two days after the surgery. A total 1mL of PDRN was injected along the suture line at distance of 1cm in each session.
  Interventions: Procedure: Polydeoxyribonucleotide (PDRN)
- Control group (No Intervention): The participants in control group were left untreated.

INTERVENTIONS:
Procedure: Polydeoxyribonucleotide (PDRN) — A total 1mL of PDRN was injected along the suture line at distance of 1cm in one day and two days after the surgery.
  Arms: PDRN injected group

SUMMARY:
The investigators aimed to evaluate the efficacy of PDRN administration in early wound healing phase on prevention of post-operative scars after open thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

• Participants who underwent open thyroidectomy between February 2019 and March 2021 at the Thyroid Cancer Center, Department of otorhinolaryngology, Seoul National University Bundang Hospital

Exclusion Criteria:

* age younger than 20 years or older than 60 years
* history of keloid development
* requirement for modified radical neck dissection
* previous neck surgery
* current pregnancy or breast feeding
* allergy to PDRN
* taking medications that may affect inflammation and would healing such as isotretinoin, anti-cancer drugs, high dose corticosteroids, and anticoagulants
* uncontrolled medical diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
modified Vancouver Scar Scale (0 normal skin~15 worst) at the 3-month follow-up | at 3 months
  modified Vancouver Scar Scale (0 normal skin~15 worst)

SECONDARY OUTCOMES:
Subjective symptoms at the 3-month follow-up | at 3 months
  Pain and itching were assessed using a visual analog scale (VAS) ranged from 0 (no) to 10 (worst).
Erythema and pigmentation at the 3-month follow-up | at 3 months
  Erythema Index (EI, arbitrary unit) and the Melanin Index (MI,arbitrary unit)
Scar Height (mm) at the 3-month follow-up | at 3 months
  3D images of the scars were acquired with an Antera 3D® camera (Miravex Limited, Dublin, Ireland)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Won Shin, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No